CLINICAL TRIAL: NCT05630872
Title: Pharmacokinetics and Safety of Double-dose Dolutegravir When Used With Rifapentine for HIV-associated Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ViiV Healthcare (Industry); Mylan Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5406
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: HIV-associated Tuberculosis
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adults with HIV and newly diagnosed DS-TB not currently on ART (Experimental): Participants will receive daily rifapentine-moxifloxacin plus isoniazid and pyrazinamide for 8 weeks followed by daily rifapentine-moxifloxacin plus isoniazid for 9 weeks (referred to as 2HPZM/2HPM) for anti-tuberculosis (anti-TB) therapy at study entry.
  DTG-based ART at 50 mg twice daily (BID) will be started after 6 weeks of TB therapy and will be continued for 2 weeks after completion of TB therapy.
  Two weeks after completion of TB therapy DTG will be reduced to standard dose 50 mg once daily (QD).
  Interventions: Drug: Dolutegravir (DTG) 50 mg orally BID (~12 hours apart) plus TDF/3TC; Drug: DTG 50 mg orally QD plus TDF/3TC; Drug: 2HPZM; Drug: 2HPM

INTERVENTIONS:
Drug: Dolutegravir (DTG) 50 mg orally BID (~12 hours apart) plus TDF/3TC — Dolutegravir (DTG) 50 mg orally BID (~12 hours apart) plus TDF/3TC, from study week 6 until 2 weeks after completion of TB treatment: Morning dose DTG 50 mg QD plus TDF/3TC from study-supplied ARV regimen. Evening dose: DTG 50 mg orally QD from study-supplied source.
Drug: DTG 50 mg orally QD plus TDF/3TC — DTG 50 mg orally QD plus TDF/3TC from two weeks after completion of TB treatment to end of study (week 48).
Drug: 2HPZM — Daily rifapentine-moxifloxacin plus isoniazid and pyrazinamide regimen
Drug: 2HPM — Daily rifapentine-moxifloxacin plus isoniazid regimen

SUMMARY:
A5406 hypothesizes that dolutegravir (DTG) 50 mg taken twice daily will provide adequate exposures to maintain viral suppression when dosed with rifapentine (RPT) 1200 mg for HIV-associated TB.

DETAILED DESCRIPTION:
This is an open-label, single arm, phase II, multicenter PK study to investigate the effect of daily RPT 1200 mg on DTG exposure in participants with HIV-associated TB. Adults with HIV with newly diagnosed DS-TB who are not currently on ART will be recruited around the time of DS TB diagnosis. At study entry, the 2HPZM/2HPM regimen will be initiated for anti-tuberculosis (anti-TB) therapy and continued for 17 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals ≥18 years of age at study entry.
2. Weight ≥40 kg.
3. Body mass index (BMI) >18.5 kg/m2.
4. Ability and willingness of participant or legal guardian/representative to provide informed consent.
5. Documentation of HIV-1 status.
6. CD4+ cell count ≥100 cells/mm3 obtained within 30 days prior to study entry at any network-approved non-US laboratory that is IQA certified.
7. ART-naïve or not on ART for 12 consecutive weeks prior to TB diagnosis.
8. Willingness and eligibility to start DTG-based ART at 6 weeks, with a window of ±1 week, after starting TB treatment, with no intention to change ART for the duration of the study.
9. Documentation of pulmonary TB.
10. Willingness to start 2HPZM/2HPM therapy for DS-TB.
11. The following laboratory values obtained within 30 days prior to study entry:

    * Absolute neutrophil count (ANC) >750 cells/mm3
    * Hemoglobin ≥7.4 g/dL
    * Platelet count ≥50,000/mm3
    * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) <2.5 X the upper limit of normal (ULN)
    * Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) <2.5 x ULN
    * Total bilirubin ≤1.5 x ULN
    * Creatinine <1.3 x ULN
12. For participants who can become pregnant, negative serum or urine pregnancy test at screening within 30 days prior to entry and within 48 hours prior to entry.
13. Participants who can become pregnant must agree not to participate in the conception process and if participating in sexual activity that could lead to pregnancy, must agree to use one reliable nonhormonal method of contraception.
14. Documentation of Karnofsky performance score ≥50 within 30 days prior to entry.

Exclusion Criteria:

1. Breastfeeding, pregnant, or plans to become pregnant.
2. Known allergy/sensitivity or any hypersensitivity to components of the study drugs, or their formulations.
3. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
4. Requirement for ongoing use of drugs that are known to have significant drug-drug interactions with DTG or RPT.
5. Known history of acute intermittent porphyria.
6. Previous treatment for active TB disease.
7. More than 5 days of treatment directed against active TB for the current TB episode preceding study entry.
8. At the time of study entry, documentation of an M. tuberculosis isolate from the current or previous treatment episode known to be resistant to RIF or INH.
9. Known history of prolonged QT syndrome.
10. Known cirrhosis, a history of decompensated liver disease (ascites, hepatic encephalopathy, or esophageal varices).
11. Documentation of severe opportunistic infections, in the opinion of the site investigator, within 3 months of study entry.
12. Documentation of severe extra-pulmonary TB (e.g., meningitis, osteomyelitis, disseminated TB) at the time of screening.
13. Acute gout at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Model-simulated 5th percentile and corresponding 95% confidence interval of DTG minimum concentrations (Cmin) at 50 mg BID when co-administered with daily RPT 1200 mg plus HZM | 48 Weeks

SECONDARY OUTCOMES:
DTG minimum concentration (Cmin) | 48 Weeks
  Model-derived participant- and week-specific estimate of DTG Cmin
DTG minimum concentration (Cmax) | 48 Weeks
  Model-derived participant- and week-specific estimate of DTG Cmax
DTG area under the concentration-time curve (AUC0-24) | 48 Weeks
  Model-derived participant- and week-specific estimate of DTG AUC0-24
Number of participants who experience Grade 3 or higher AEs | Weeks 6-17
Number of participants who have a diagnosis of rifamycin hypersensitivity | Weeks 6-17
Number of participants who experience ALT ≥3xULN with symptoms/jaundice or ALT ≥5xULN | Weeks 6-17
Number of participants who prematurely discontinue study drugs DTG and/or RPT | Weeks 6-17
Proportion of participants with HIV-1 viral load below 50 copies/mL | Weeks 10, 14, 21, and 30

CONTACTS AND LOCATIONS:
Locations (4):
- South Africa (3):
  - University of Cape Town Lung Institute (UCTLI) CRS (Site # 31792), Mowbray, Cape Town, Western Cape
  - Durban International CRS (Site # 11201), Westridge, Durban RSA
  - South African Tuberculosis Vaccine Initiative (SATVI) CRS (Site # 31793), Worcester, Western Province
- Thai Red Cross AIDS Research Centre (TRC-ARC) CRS (Site # 31802), Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.